### HOSPITAL FOR SPECIAL SURGERY

535 East 70<sup>th</sup> Street New York, NY 10021

# INFORMED CONSENT TO PARTICIPATE IN RESEARCH

TITLE: The Combination of Adductor Canal Block and Peri-Articular Injection with an Accelerated Rehabilitation Protocol. A Novel Technique for Patients Undergoing Total Knee Replacement

PROTOCOL NO.: 2014-018

SPONSOR: HSS Department of Anesthesiology, HSS Department of Rehabilitation, Adult Reconstruction and Joint Replacement Division

INVESTIGATOR: Enrique Goytizolo, MD

SITE(S): Hospital for Special Surgery

### STUDY-RELATED PHONE NUMBER(S):

(212) 797-8676: Enrique Goytizolo, MD Principal Investigator

(212) 774-7022: Katie (Phuong Dinh) Mac, BA Research Assistant

(212) 774-7377: Jennifer Cheng, PhD Research Associate

IRB #: 2014-018


You are being asked to take part in a research study conducted by Hospital for Special Surgery (HSS). You are being asked to participate in this study because you are to undergo total knee replacement surgery by Dr. Alexiades, Dr. Mayman, Dr. Padgett, Dr. Amar Ranawat, Dr. Su, or Dr. Westrich.

You will still be responsible for the cost of your medical care just as you would be if you were not part of this study. For example, any co-pays, deductibles, and co-insurance associated with your medical care.

This document provides you with information about this study. After reading this document, any questions you may have will be answered. You may take home a copy of this document to consider or discuss with family and friends before making your decision.

A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Form 10 - ICF Document (Template Version 2/14/13)

IRB Administrative Use Only

Hospital for Special Surgery Institutional Review Board Approval 7/14/2016 Thru 3/24/2017

Review Board Ap

### 1. WHY IS THIS STUDY BEING DONE?

Relieving post-operative pain is extremely important to orthopedic surgeons and anesthesiologists at HSS. The purpose of this study is to compare the effectiveness of two methods of pain control along with an accelerated physical therapy protocol in aiding the achievement of rehabilitation milestones. The two pain control methods include: (1) peri-articular injections during the surgery and (2) peri-articular injections during the surgery and a peripheral nerve block. The peri-articular injections are performed by your surgeon and are injections of pain medicine around the knee. The nerve block (injection of local anesthetic, numbing medicine, near a nerve leading to the knee) being investigated in this study is the adductor canal block. The adductor canal block has been shown to decrease pain and morphine use and preserve quadriceps strength post total knee replacement. Your overall participation will continue over the course of your hospital stay at the Hospital for Special Surgery.

## 2. WHAT WILL YOUR PARTICIPATION REQUIRE?

If you decide to be in this study, the following routine and/or experimental procedures will be performed:

| Study | Surveys / | Randomization | Surgery | Physical | Physical | Physical |
|---|---|---|---|---|---|---|
| Visit # | Questionnaires | | | Therapist | Therapist | Therapist |
| | | | | Visit #1 | Visit #2 | Visit #3 |
| Holding | X | X | SOC | | | |
| Area | | | | | | |
| PACU | X | | | SOC | | |
| POD 1 | X | | | SOC | X (until | X (until |
| | | | | | Rehab | Rehab |
| | | | | | goals are | goals are |
| | | | | | met) | met) |
| POD 2 | X | | | SOC | X (until | X (until |
| | | | | | Rehab | Rehab |
| | | | | | goals are | goals are |
| | | | | | met) | met) |

### X= Research procedures

SOC= Standard of care (care you would receive if you were not participating in this study)

This study will select your treatment by chance. You will be assigned at random to one or more study groups:

## Group 1 - Peri-articular Injection group

A spinal anesthetic with 0.5% bupivacaine (10 or 12.5mL) will be performed. The surgeon will perform the periarticular injections. The deep injection will consist of bupivacaine 0.5% with epinephrine, 30cc; morphine, 8 mg/ml, 1 cc; methylprednisolone, 40 mg/ml, 1 ml; cefazolin, 500 mg in 10 ml; normal saline, 22cc. The superficial injection will be 20 ml 0.25% bupivacaine. Patients will also be given 2 mg of intravenous decadron


IRB Administrative Use Only

## Group 2 – Peri-articular + Adductor Canal Block group

In addition to the above peri-articular injection protocol, patients will receive an adductor canal block: 15 cc of Bupivacaine 0.25% with 2 mg of Preservative free Dexamethasone.

The randomization process is comparable to (or similar to) the flip of a coin. It is not known if any treatment you receive will benefit you. It is hoped the knowledge gained will benefit others in the future. You, as well as the research, nursing, physical therapist, and acute pain staff will be blinded as to which study group you are in. However, your anesthesiologist will not be blinded.

You and/or your insurance will be responsible for any costs of all procedures performed that are standard of care, that is, care that you would receive even if you were not in this study.

A total of 114 subjects will participate in this study at HSS.

Your participation will involve a total of 6 study visits. Most visits are expected to last 5-10 minutes.

# 3. WHAT ADVERSE (BAD) EFFECTS CAN HAPPEN FROM BEING IN THE STUDY? WHAT RISKS ARE KNOWN ABOUT THE STUDY DRUG/STUDY DEVICE?

The known effects, discomforts and foreseeable risks of physical, psychological, sociological, or other harm which you may reasonably expect to occur from being in this study are:

- Adductor Canal Block: One group will receive the adductor canal block. This will be an injection of local anesthetic near the saphenous nerve with ultrasound guidance. It is a possibility that the nerve may become irritated or injured during the injection. Your anesthesiologist will talk with you more about this procedure.
- Peri-articular Injection: Both groups will receive the peri-articular injection. This is an injection performed near the knee joint by your surgeon. The injection is a combination of local anesthetic and other medications hoped to reduce pain and side effects. It is possible that the tissue near the knee may become irritated or injured with the injection.
- Opioids: Opioids are given to both groups pre operatively and are used for pain control after total knee replacement. Sometimes nausea, vomiting, itching, sedation and confusion, and constipation can occur.
- Other Medications: Meloxicam (an oral non-steroidal anti-inflammatory drug) is used in both groups. It is standard of care at HSS for total joint replacements and is thought to reduce pain and improve mobility. Meloxicam is rarely associated with kidney problems. Steroids are given in both groups. Usually significant side effects do not occur with a single dose, but a short term rise in blood sugar is possible.

Participation in this research involves the potential risk of a breach of confidentiality to your stored health information. HSS tries to minimize those risks by (i) removing some direct identifiers from stored information [(i.e., names, social security numbers, medical record numbers); (ii) securing, in a separate location, and limiting access to information that would identify you; and (iii) limiting access to information stored to HSS investigators.


IRB Administrative Use Only

There may be risks or side effects that are unknown at this time. If we learn about new risks that may affect your willingness to continue your participation, we will make you aware of them and you will be asked to re-consent to continue your participate in the study.

Your condition may not get better from being in this study. Your condition may or may not get worse from being in this study.

### 4. WHAT BENEFIT CAN YOU EXPECT?

All patients participating in the study will receive an accelerated physical therapy program postoperatively, at no cost to you.

If you are in the group receiving peri-articular injections (50% chance) you may or may not receive any additional benefit. If you are in the group receiving peri-articular injections and the adductor canal block (50% chance) you may or may not experience less pain. If you experience less pain then you may reduce your opioid consumption. Reduced opioid consumption could lead to fewer opioid related side effects. Such side effects include constipation, nausea, vomiting, sedation, sleepiness, difficulty concentrating, difficulty urinating, and dry mouth.

### 5. COST

Those research procedures listed in Section 2 will be covered by the study and will not be your financial responsibility.

As indicated in Section 2, those costs which are considered Standard of Care for your treatment here at Hospital for Special Surgery will be your/or your insurance's responsibility. You will be responsible for any co-pays, deductibles, and co-insurance associated with your medical care, just as you would be for any costs billed to your health insurance outside of this study. You will also be financially responsible for any medical care costs not covered by your health insurance.

HSS is committed to providing financial assistance when financially warranted and consistent with its resources, regardless of age, gender, religion, race or sexual orientation. So if you do not have health insurance, or if your health insurance does not pay for your medical care, you may seek financial assistance from HSS. Eligibility determinations are made on a case-by-case basis in accordance with HSS's financial assistance policy. You will be responsible for any costs not covered by financial assistance, which could be all of the costs (if HSS determines that you are not eligible for financial assistance) or some of the costs (if financial assistance awarded by HSS does not cover all of the costs). For more information about the Financial Assistance

Program or to request a Financial Assistance Application call (212) 606-1505 to speak with a Financial Assistance Counselor or you can visit the following site:

http://www.hss.edu/patient-financial-assistance-notice.asp.

### 6. PREGNANCY

Due to inherent risks, HSS policy prevents women who are pregnant or nursing a child from receiving the type of surgery or procedure needed to qualify for this research study. So if you are currently pregnant or nursing a child, you may not participate in this study.


IRB Administrative Use Only

Hospital for Special Surgery Institutional Review Board Approval 7/14/2016 Thru 3/24/2017


### 7. PAYMENT FOR PARTICIPATION

You will not be paid for your participation in this study.

### 8. COMMERCIAL ISSUES: YOUR RIGHTS IN THE RESULTS OF THE STUDY

There are no plans to compensate you for the use of the findings of this study, or any of the information or biologic materials (such as blood or tissue) collected from you during the study, even if they are used to develop or make a commercial product (such as a drug, device, biologic substance, or test).

# 9. ALTERNATIVES: WHAT OTHER TREATMENT IS AVAILABLE IF YOU DON'T WANT TO BE IN THE STUDY?

You do not have to participate in this study to receive treatment for your condition.

# 10. WHO WILL BE ABLE TO SEE YOUR RECORDS AND PERSONAL INFORMATION AND KNOW THAT YOU ARE IN THE STUDY?

Federal regulations give you certain rights related to your health information. These include the right to know who will be able to see your information and why they will be able to see it. The study doctor must obtain your authorization (permission) to use or give out any health information that might identify you.

# What information may be used or given to others?

If you choose to be in the study, the study doctor will get personal information about you. The information might identify you. The study doctor may also get information about your health including:

- Medical and research records
- Records about phone calls
- Records about your study visits
- Records of physical exams
- Laboratory, x-ray, and other test results
- Questionnaires
- Records about any study device you received

# Who may use, disclose, or receive my information?

The following person(s) class(es) of persons, and/or organization(s) may use, disclose, or receive my information:

- The Principal Investigator and other Investigators for this study, including your study doctor.
- The research coordinator, research nurses, and other members of the HSS research team working on this study.


IRB Administrative Use Only


- Every research site for this study, including Hospital for Special Surgery and its affiliates, New York-Presbyterian Hospital, and Memorial Sloan-Kettering Cancer Center. This includes the research staff and medical staff at each institution.
- The Patient Advocate or Research Ombudsman at these institutions.
- Staff members of HSS responsible for administering clinical trials and other research activities
- Any laboratories and other individuals and organizations that analyze your health information for this study.
- Any health care provider that you have used in the past or may use up to the time this study ends.
- The United States Food and Drug Administration (FDA), the federal Office for Human Research Protections (OHRP), any federal agency that provides support for this study, and any federal, state, or local agency responsible for overseeing HSS, the study doctor, or any other member of the HSS research team involved in this study.
- The members and staff of the affiliated Institutional Review Boards (IRBs) at HSS, New York-Presbyterian Hospital, and Memorial Sloan-Kettering Cancer Center. An IRB is a committee of health care providers, community representatives, and others that initially approves and periodically reviews biomedical and behavioral research that involves human subjects in order to protect the rights, safety and welfare of study participants.
- Data Safety Monitoring Boards and others authorized to monitor the conduct of this study for safety or quality assurance, for example a Clinical Events Committee.

# Why will this information be used and/or given to others?

Your health information may be given to others to carry out this study. The research staff will analyze and evaluate the results of this study.

Your health information may be given to the FDA. It may also be given to governmental agencies in other countries. Your information may also be used to meet the reporting requirements of governmental agencies.

The results of this study may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

## What if I decide not to give permission to use and give out my health information?

By signing this informed consent form, you are giving permission to use and give out your health information as described above. If you refuse to give permission, you cannot be in this study.

## May I review or copy the information obtained from me or created about me?

You have the right, in accordance with Hospital policy and applicable law, to review and copy your health information that is created or obtained in the course of this study. However, if you decide to be in this study and sign this informed consent form, you will not be able to look at or copy your information until after the study is completed if doing so would impact the validity of


IRB Administrative Use Only

the study (for example, if the study is "blinded" so that during the study you will not know what treatment or other intervention you are receiving).

# May I revoke (take back) my permission?

Yes. Your permission will never expire unless you revoke it. To revoke your permission, you must write to the study doctor at Hospital for Special Surgery, 535 East 70<sup>th</sup> Street, New York, NY 10021.

You may revoke your permission to use and disclose your health information at any time. If you revoke your permission, you cannot continue to participate in this study.

After you revoke your permission, no new health information that might identify you will be gathered. Information that has already been gathered may still be used and given to others. This would be done if the information is needed for this study to be reliable.

<u>Is my health information protected after it has been given to others?</u>

Some persons who receive your health information may not be required to protect it, and they may share your information with others without your permission, if permitted by laws governing them. Therefore, there is a risk that your information will be released to others without your permission.

## 11. CONFLICT OF INTEREST NOTIFICATION

HSS is concerned about possible conflicts of interest in research, and has policies that require all investigators and senior research staff to report to HSS significant financial interests (such as stock ownership, royalty payments, and consulting agreements) and relationships (such as membership on a scientific advisory board) that are related to their research studies. When an investigator reports a significant financial interest or relationship that relates to one of his/her studies, HSS's Conflict of Interest Committee for Research reviews the information to evaluate the risk that the interest or relationship might influence how the investigator conducts the study or interprets the results of the study. HSS may also take steps to minimize that risk.

| The Conflict of Interest Committee for Research has determined that there are no conflicts of interest associated with this study. |
|---|
| The Conflict of Interest Committee for Research has determined that there is a potential conflict of interest associated with this study. Please read the information below carefully. |

### 12. VOLUNTARY PARTICIPATION/WITHDRAWAL

Your decision to take part in this study is completely voluntary. You are free to choose not to take part in the study and may change your mind and withdraw at any time. Your relationship with physicians at HSS and your medical care at HSS, now or in the future, will not be affected


IRB Administrative Use Only

Hospital for Special Surgery Institutional Review Board Approval 7/14/2016 Thru 3/24/2017

**** 

in any way if you withdraw or refuse to participate. You will not lose any benefits to which you are otherwise entitled.

The study doctor and/or the sponsor may terminate your participation in this study at any time without your consent if, in their judgment, it is inadvisable for you to continue.

### 13. COMPENSATION FOR INJURY

If you are injured as a result of participating in this study, the study doctor, other members of the research team, or other HSS professional medical staff will provide you with emergency medical treatment (or arrange to have such treatment provided to you), and will assist you in obtaining appropriate follow-up medical treatment. However, there is no plan to routinely provide compensation for additional medical care or other costs.

Your health insurance may or may not pay for treatment of injuries as a result of your participation in this study.

### 14. SOURCE OF FUNDING

Funding for this study will be provided by the HSS Department of Anesthesiology, HSS Department of Rehabilitation, and the Adult Reconstruction and Joint Replacement division.

### 15. QUESTIONS

If you have any additional questions later on, or if you wish to report a medical problem that may be related to this study, Dr. Enrique Goytizolo can be reached at 212-797-8676 during office hours.

If you have any questions about your rights as a participant in this study or any questions about your participation that you would like to ask an institutional representative who is not part of this study, you can call the Manager of the HSS Institutional Review Board at (212) 774-7154.

If you would like to have more information about the Hospital's financial disclosure review process in general, or in regard to this study, you may contact the Hospital's Office of Legal Affairs at (212) 606-1592. You may also ask the Hospital's patient advocate at (212) 774-2403, to arrange for you to have this information.

Do not sign this consent form unless you have had a chance to ask questions and have received satisfactory answers to all of your questions.


IRB Administrative Use Only


# Agreement to Participate: Witnessing and Signature

To be in this study, you or your legal representative must sign the next page of this informed consent form. By signing the next page, you are voluntarily agreeing to be in this study at HSS.

Before signing, you should be sure of the following:

- You have read all of the information in this "Informed Consent to Participate in Research" form (or had it read to you).
- You have discussed the implications of your being in this study with your doctor, your study doctor and/or the study coordinator.
- You have had the chance to ask questions about this study.
- You received answers to your questions.
- If you did not understand any of the answers, you asked the study doctor or the study coordinator to explain them to you.
- The information given to you is based on what is now known about the study drug(s), device(s), or procedure(s). There may be other risks or complications that are not known at this time.
- You have had time to think about the information and decide whether or not to be in the study.

| Please ch | eck one of the following: |
|-----------|--------------------------------------------------|
| | I AM NOT in another research study at this time. |
| | I AM in another research study at this time. |


IRB Administrative Use Only

If you decide to be in this study:

- You are expected to follow the study procedures.
- You are expected to provide the information needed by the study doctor, the study coordinator, nurses, or other staff members for the study.
- You will be told in a timely manner of any significant new information that may affect your willingness to stay in the study.
- You may freely choose to stop being in the study at any time.

By signing below, you are voluntarily agreeing to be in this study.

You must be given a signed copy of this informed consent form to keep for yourself.

| Print Name of Participant | Signature of Participant | Date |
|---|---|---|
| Print Name of Parent/Legal Guardian (if applicable) <sup>1</sup> | Signature of Parent/Legal Guardian | Date |
| Print Name of Person Obtaining Consent | Signature of Person Obtaining Consent | Date |

As an HSS representative, please sign here to indicate that you have given a signed copy of this informed consent form to the participant

### **NOTE TO INVESTIGATORS:**

- THE ORIGINAL OF THIS INFORMED CONSENT FORM MUST BE PLACED IN THE PARTICIPANT'S STUDY FILE.
- A SIGNED COPY OF THIS INFORMED CONSENT FORM MUST BE GIVEN TO THE PARTICIPANT.
- A COPY OF THE INFORMED CONSENT FORM MUST BE PLACED IN THE PARTICIPANT'S HOSPITAL MEDICAL RECORD IF THE PARTICIPANT IS (OR WILL BE) HOSPITALIZED AT ANY TIME DURING THE STUDY.


IRB Administrative Use Only

Hospital for Special Surgery Institutional Review Board Approval 7/14/2016 Thru 3/24/2017


<sup>&</sup>lt;sup>1</sup> The parent or legal guardian of a child participant should sign this form on behalf of the child. The signature of one parent is sufficient when the research is of minimal risk to the child, or when the research presents the prospect of direct benefit to the child. The signature of both parents is required when the research involves greater than minimal risk with no prospect of direct benefit to the child. The requirements for signature of both parents may be waived if one parent is deceased, unknown, incompetent, or not reasonably available, or when one parent has sole legal responsibility for the care and custody of the child. If the participant is a child who is capable of giving assent, the child should also sign the attached Assent Form.